CLINICAL TRIAL: NCT05745961
Title: Quantifying 18kDa TSPO Expression in the Lung in Pulmonary Artery Hypertension (PAH)
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 22HH8097
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Arterial Hypertension; Healthy
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — (methyl-(11)C)N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PAH
  Interventions: Radiation: TSPO PET scan (11C-PBR28)
- Healthy volunteer
  Interventions: Radiation: TSPO PET scan (11C-PBR28)

INTERVENTIONS:
Radiation: TSPO PET scan (11C-PBR28) — PET scan

SUMMARY:
The aim of this study is to determine whether there is an increase in the TSPO PET signal (measured with the radioligand [11C]PBR28) in the lungs of patients living with PAH relative to age matched controls. If so, TSPO PET may be a useful technique to non-invasively monitor response to therapy. To do this, we will perform 2 [11C]PBR28 PET scans. The first will quantify the total [11C]PBR28 PET signal. This signal is a combination of the specific signal (VS) and the nonspecific signal (VND). The second scan will be performed following dosing with an unlabelled TSPO ligand. By directly measuring the total [11C]PBR28 signal (scan 1) and the nonspecific [11C]PBR28 signal (scan 2) we can therefore calculate the specific [11C]PBR28 signal, and hence the amount of TSPO in the lung.

ELIGIBILITY:
Inclusion Criteria:

Able to provide written informed consent prior to any study mandated procedures.

Able to lie comfortably on back for up to 90 minutes at a time.

Fertile females (women of childbearing potential) are eligible to participate after a negative highly sensitive pregnancy test, if they are taking a highly effective method of contraception other than the oral contraceptive pill until the end of relevant systemic exposure.

Male participants who are fertile are eligible to participate if they are willing to comply with the contraceptive requirements

Exclusion Criteria:

Unable to provide informed consent and/or are non-fluent speakers of the English language

TT Genotype at the rs6971 locus

Clinically-significant renal disease (confirmed by creatinine clearance <30 ml/min per 1.73m2)

Clinically-significant liver disease (confirmed by serum transaminases >2 times than upper normal limit)

Anaemia confirmed by haemoglobin concentration <10 g/dl

Sickle cell disease or thalassaemia

History of uncontrolled systemic hypertension

Acute infection (including eye, dental, and skin infections)

Chronic inflammatory disease including HIV, and Hepatitis B

Women of childbearing potential who are pregnant or breastfeeding

Patients who have received an Investigational Medicinal Product (IMP) within 5 half-lives of the last dose of the IMP or 1 month (which ever is greater) before the baseline visit

Participation in a research study involving significant ionisation radiation within the last 3 years

Significant radiation exposure other than dental X-rays in last 1 year

Positive Allen's test.

-

Ages: 25 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: PAH patients and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
The specific and non-specific fractions of the [11C]PBR28 signal in the lungs of healthy individuals and PAH patients. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wilkins, Principal Investigator — Imperial College London
Locations (1):
- Imperial Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided